CLINICAL TRIAL: NCT06142370
Title: The Prevalence of the Linburg-Comstock Variation in Patients With Symptomatic Thumb CMC Arthritis
Brief Title: The Prevalence of the Linburg-Comstock Variation
Acronym: LCV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Russell Sage College (Other)
Collaborators: Albany Medical College (Other)
Responsible Party: Principal Investigator, Christine Mulligan, Assistant Professor, Russell Sage College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RussellSage1
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Anomaly; Hand
MeSH Terms: conditions — Hand Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive LCV (Other): A patient who tests positive by clinical exam of a LCV.
  Interventions: Other: Descriptive

INTERVENTIONS:
Other: Descriptive — The patients will be asked by the recruiting physicians to perform a clinical examination looking for the LCV, which will take a total of five seconds. This is a self-test and not part of a regular clinical examination

SUMMARY:
The purpose of this study is to explore the physical exam characteristics of patients referred to orthopedic surgeons with a diagnosis of thumb carpometacarpal (CMC) arthritis. CMC osteoarthritis of the thumb is one of the most common degenerative conditions of the hand in 11% of men and 33% of women (Gillis et al., 2011). Patients with CMC arthritis may experience pain, decreased range of motion, loss of grip and pinch strength, often limiting participation in activities of daily living (Bertozzi et al., 2014). In 1979, two physicians identified a variation of a tendinous connection in the wrist between the tip of the index finger and the tip of the thumb known as the Linburg-Comstock variation (LCV) (Linburg & Comstock, 1979). The prevalence of the LCV varies respectively from 13-66% in both males and females (Erić et al., 2019). A physical examination of patients with LCV reveals concurrent flexion of the flexor digitorum profundus to the index finger and flexor pollicis longus. The study aims to gain more insight into patients diagnosed with CMC arthritis through clinical examination for LCV to consider an association of the diagnoses.

Currently, there is no evidence surrounding patients with symptomatic CMC arthritis and LCV. The hypothesis is that there is an association between symptomatic CMC arthritis and LCV. Patients with a LCV may then be more likely to develop painful CMC arthritis.

DETAILED DESCRIPTION:
Five hundred male and female patients over the age of 35 will be recruited to participate through convenience sampling. This is a descriptive cross-sectional study of patients with a diagnosis of thumb CMC arthritis. There is no control group due to the recruitment of one patient population. Once enrolled, commitment of the participants will consist of one time during their regular office visit. The patients will be asked by the recruiting physicians to perform a clinical examination looking for the LCV, which will take a total of five seconds. This is a self-test and not part of a regular clinical examination.

Subjects meeting the inclusion criteria will be consented during office clinic visit with Dr. Michael Mulligan, Dr. Richard Uhl, Dr. Patrick Marinello, Dr. Andrew Morse, Dr. George Zanaros, Dr.

Whipple and Dr. David Quinn. The descriptive study will collect demographic data, and dichotomous data indicating whether a patient has the variation or does not have the variation, and if the variation is present in one hand or both hands. The study will take place at the Bone and Joint Center at 1365 Washington Avenue, Albany New York, and satellite offices in Guilderland, Clifton Park, Malta, Saratoga, Schenectady and Catskill. Data will be collected for up to two years. There are no risks to patients enrolled in the study, as the test involves asking the patient to simply bend the tip of their thumb. Documentation of the variation is not usually noted in the chart. Therefore, the physicians involved in the study will be asked to include the findings of the variation in their documentation. The patients will be informed during clinical examination if they have a LCV. There is no compensation to participants for enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female

  * Over the age of 35
  * Under the age of 89
  * Diagnosis of thumb CMC arthritis, ICD-10 code M19.12
  * Initial non-surgical intervention for thumb CMC arthritis

Exclusion Criteria:

* Under the age of 35
* Over the age of 89
* Prisoners

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
LCV | 10 seconds
  A positive or negative clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Chris Mulligan, Principal Investigator — Russell Sage College
Locations (1):
- The Bone and Joint Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided